CLINICAL TRIAL: NCT03064815
Title: Prevalence of Small Bowel Inflammatory Crohn's Disease Lesions in Patients With Spondyloarthropathies (SpA): A Prospective Capsule Endoscopy-Based Study
Brief Title: The SpACE Study - Small Bowel Crohn's Disease and Spondyloarthropathies
Acronym: SpACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: AbbVie (Industry); Prometheus Laboratories (Industry)
Responsible Party: Principal Investigator, Ernest Seidman, Director of Research in IBD at McGill University, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GEN-08-053
Record Dates: First submitted 2017-02-10; First posted 2017-02-27 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Spondyloarthropathy; Crohn Disease
MeSH Terms: conditions — Spondylarthropathies; Crohn Disease | interventions — Capsule Endoscopy; Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spondylarthropathies with GI symptoms (Experimental): Subjects in this arm will have spondylarthropathies and gastrointestinal symptoms and will undergo a colonoscopy, videocapsule endoscopy, biomarker testing (PROMETHEUS® IBD sgi Diagnostic™ and fecal calprotectin)
  Interventions: Device: Videocapsule endoscopy; Procedure: colonoscopy; Diagnostic Test: PROMETHEUS® IBD sgi Diagnostic™; Diagnostic Test: Fecal calprotectin
- Spondylarthropathies without GI symptoms (Experimental): Subjects in this arm will have spondylarthropathies without gastrointestinal symptoms and will undergo a colonoscopy, videocapsule endoscopy, biomarker testing (PROMETHEUS® IBD sgi Diagnostic™ and fecal calprotectin)
  Interventions: Device: Videocapsule endoscopy; Procedure: colonoscopy; Diagnostic Test: PROMETHEUS® IBD sgi Diagnostic™; Diagnostic Test: Fecal calprotectin

INTERVENTIONS:
Device: Videocapsule endoscopy — Capsule endoscopy is a procedure that uses a tiny wireless camera to take pictures of your digestive tract. A capsule endoscopy camera sits inside a vitamin-size capsule you swallow. As the capsule travels through your digestive tract, the camera takes thousands of pictures that are transmitted to a recorder you wear on a belt around your waist.
  Capsule endoscopy helps doctors see inside your small intestine - an area that isn't easily reached with more-traditional endoscopy procedures.
  Other Names: Capsule endoscopy
Procedure: colonoscopy — Colonoscopy is a test that allows your doctor to look at the inner lining of your large intestine (rectum and colon). He or she uses a thin, flexible tube called a colonoscope to look at the colon.
Diagnostic Test: PROMETHEUS® IBD sgi Diagnostic™ — This test combines serologic, genetic, and inflammation markers in a proprietary Smart Diagnostic Algorithm to provide added IBD diagnostic clarity. This test helps physicians differentiate IBD vs. non-IBD and CD vs. UC in one comprehensive blood test.
Diagnostic Test: Fecal calprotectin — A stool test to measure inflammation in the gut.

SUMMARY:
Inflammatory bowel disease is clinically associated with spondylarthropathies in 5-15% of cases. Protocol colonoscopic assessment demonstrated asymptomatic inflammation characteristic of Crohn's disease in up to 1/3 of SpA patients. Videocapsule endoscopy is a superior diagnostic tool to detect small bowel mucosal pathology. However, it has been infrequently used to evaluate bowel inflammation in spondylarthropathies. This study compared the accuracy of videocapsule endoscopy to standard ileocolonoscopy for the detection of inflammatory bowel lesions in patients with spondylarthropathies, and to describe the clinical and laboratory predictors of small bowel inflammation in this cohort.

DETAILED DESCRIPTION:
The link between chronic inflammatory bowel disease and arthritis is well established. IBD is associated with 3 patterns of arthritis (1), one of which is spondylarthropathy (2). spondylarthropathies is not uncommon, with 3-6% of patients with IBD affected, while radiologic sacroileitis is evident in up to 18% of patients. SpA associated with IBD differs from that of idiopathic ankylosing spondylitis in that the prevalence of HLA-B27, although high (20-40%), is significantly lower than in typical AS, where its prevalence is characteristically 90%. Both inflammatory bowel disease and spondylarthropathies show familial clustering and may coexist. Idiopathic ankolysing spondylitis and ankolysing spondylitis usually occurs without overt signs of intestinal inflammation. However, ileocolonoscopy studies have shown a high prevalence (30-44%) of asymptomatic inflammation of the terminal ileum. The nature of this inflammation is highly characteristic of Crohn's disease. Among spondyloarthropathies patients with subclinical inflammation, only 6% were reported to eventually develop clinically apparent inflammatory bowel disease. A more recent review of endoscopy-based studies detected Crohn's disease more frequently, in 18-48 % of patients with spondyloarthropathies and in 5-11% of ankolysing spondylitis.. However, conventional endoscopic and radiological techniques are limited in their capacity to investigate the entire small bowel, and could easily miss significant mucosal lesions due to Crohn's disease.

Capsule endoscopy has been shown to be superior to conventional diagnostic techniques for the investigation of suspected Crohn's disease. The primary objective of this study is to demonstrate that this safe, non-invasive technique will reveal unidentified small bowel lesions in asymptomatic subjects with spondylarthropathies or ankolysing spondylitis more reliably than ileo-colonoscopy with biopsies.

Clinical implications: Spondylarthropathies, ankolysing spondylitis and inflammatory bowel disease are clinically, genetically and pathologically linked. Anti-tumor necrosis factor agents, including Adalimumab, Etanercept and Infliximab, are all efficacious and cost-effective in treating spondylarthropathies and ankolysing spondylitis. Since only some anti-TNF molecules are highly effective for both Crohn's disease and spondylarthropathies and related arthropathies, the present study ideally would lead to a change in general therapeutic practice, leading to wider use of molecules with a wide scope of therapeutic success.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients with spondylarthropathies or ankolysiing spondylitis, according to European Ppondyloarthropathy Study Group criteria or New York Criteria:

Exclusion Criteria:

* Patients having been or are currently exposed to an anti-tumour necrotic factor treatment (Adalimumab or Infliximab). Patients treated with anti-tumour necrotic factor receptor antibodies (Etanercept) are not excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2009-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of subjects with ankolysing spondylitis, with or without gastrointestinal symptoms, diagnosed with small bowel Crohn's disease via videocapsule endoscopy. | 2 years
  Accuracy of diagnosing small bowel Crohn's disease in patients with ankolysing spondylitis.

SECONDARY OUTCOMES:
Number of subjects with ankolysing spondylitis diagnosed with small bowel Crohn's disease compared to same subjects serological biomarkers and colonoscopy results. | 2 years
  Determine how accurate capsule endoscopy is in diagnosing small bowel crohn's disease in patients with ankolysing spondylitis.as compared to serology, fecal biomarkers and serological tests
Number of subjects with ankolysing spondylitis diagnosed with small bowel Crohn's disease whose treatment changed as a result of the diagnosis of small bowel Crohn's disease. | 2 years
  Evaluate whether the capsule findings alter or impact management of ankolysing spondylitis patients with small bowel Crohn's disease.
Determine whether genetic polymorphisms or human leukocyte antigen haplotypes are associated with concurrent spondylarthropathies and inflammatory bowel disease. | 1 yr post sample collection
  Genetic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Seidman, MD, Principal Investigator — Research Institute of the MUHC; Michael Starr, MD, Principal Investigator — Research Institute of the MUHC
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Patients will be told of the results of all blood work and diagnostic tests. Data will be presented at scientific conferences as well as published in scientific journals.
Supporting Information: Study Protocol, CSR
Time Frame: As data is compiled and assessed it will be shared via abstracts, presentations and manuscripts.